CLINICAL TRIAL: NCT00235898
Title: A Multi-Center, Open Label, Parallel Group, Randomised, Phase IIB Clinical Trial to Evaluate the Safety and Efficacy of CoFactor and 5-FU Versus Leucovorin and 5-FU in Subjects With Metastatic Colorectal Carcinoma
Brief Title: Clinical Trial in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mast Therapeutics, Inc. (Industry)
Responsible Party: Joachim Schupp, MD, Adventrx Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-CoFactor
Record Dates: First submitted 2005-10-06; First posted 2005-10-12 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Colon Cancer; Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — 5,11-methenyltetrahydrohomofolate; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): CoFactor, 5-FU
  Interventions: Drug: CoFactor; Drug: 5-FU
- 2 (Active Comparator): Leucovorin, 5-FU
  Interventions: Drug: 5-FU; Drug: Leucovorin

INTERVENTIONS:
Drug: CoFactor
  Other Names: ANX-510
  Arms: 1
Drug: 5-FU
  Other Names: 5-Fluorouracil
Drug: Leucovorin
  Arms: 2

SUMMARY:
The objective of this trial is to compare efficacy and safety of CoFactor and 5-fluorouracil (5-FU) versus leucovorin and 5-FU in treatment of metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have surgically incurable, confirmed metastatic colon or rectal adenocarcinoma.
* Be male or non-pregnant, non-lactating female subjects ≥ 18 years of age.
* If female, and of childbearing potential, agree to use adequate contraception (as deemed by the investigator) throughout their participation in this study and for 30 days after discontinuation of study medication.
* If, female of childbearing potential, have a negative pregnancy test prior to the start of the study.
* Have a life expectancy of at least 6 months.
* Have radiologically or clinically measurable disease for response assessment. Presence of ascites or pleural effusion(s) are not acceptable as single sites of response assessment, but may be present if dimensional or other discrete measurable disease is present for evaluation.
* Have an ECOG Performance Level of 0-2 (or Karnofsky of 100-70). A lower ECOG or Karnofsky is acceptable only if clearly due to non-oncologic conditions (e.g., prior paraplegia from polio).
* Have had no prior chemotherapy for established, metastatic disease. (Subjects may have received adjuvant chemotherapy with fluoropyrimidine therapy).
* Have at least 6 months elapsed since prior adjuvant 5-FU or CPT-11 therapy, or Mitomycin C or nitrosourea therapy.
* Have had at least an 8 week interval since any prior radiation therapy or 4 weeks since any major surgery.
* Have recovered from any toxicities resulting from prior therapies (except for alopecia).
* Adequate renal, bone marrow, liver function defined as serum creatinine less than 1.5 times the upper limit of normal, serum bilirubin less than 2 times the upper limit of normal, ANC greater than 1.5 x 109/L, Platelet count greater than 90 x 109/L, SGOT (AST) and SGPT (ALT) less than 3 times the upper limit of normal.

Exclusion Criteria:

* Failure by the subject or the subject's legal representative to sign the Informed Consent.
* An inability to obtain Informed Consent because of psychiatric or complex medical problems.
* Have concurrent infection including diagnoses of FUO or evidence of possible central line sepsis (subjects must be afebrile at the start of therapy).
* Have unstable oncologic emergency syndromes: superior vena cava (SVC) syndrome, rising bilirubin needing stent placement, spinal cord compression, progressive brain metastases, active bleeding, hypercalcemia, etc.
* Have unstable medical conditions such as acute coronary syndrome, cardio-vascular accident within the previous 12 months (such as transient ischemic attacks, accelerated hypertension), etc.
* Have cerebellar neurologic syndromes such as Parkinson's disease, multiple sclerosis, and amyotonia.
* Have a known intolerance to fluoropyrimidine (5-FU, Capecitabine, Floxuridine, UFT) therapy (dihydropyrimidine dehydrogenase deficiency).
* Patients with vomiting, diarrhea, or nausea of grade greater than 1.
* Received any investigational drug or agent/procedure, i.e. participation in another trial within 4 weeks before beginning treatment with study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2005-05; Primary Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Cassidy, MD, Principal Investigator — Beatson Oncology Centre
Locations (30):
- India (10):
  - Global Hospital, Hyderabad, Andhra Pradesh
  - Department of Medical Oncology, Nizam's Institute of Medical Sciences, Hyderabad, Andhra Pradesh
  - Kasturba Medical College, Mangalore, Attavar
  - Department of Medical Oncology, Deenanath Mangeshkar Hospital and Research Centre, Pune, Erandawane
  - Department of Medical Oncology, Kidwai Memorial Institute of Oncology, Bangalore, Karnataka
  - Department of Oncology, Christian Medical College, Vellore, Tamil Nadu
  - Manipal Hospital, Bangalore
  - SMS Medical College Hospital, Jaipur
  - Department of Medical Oncology, Dayanad Medical College and Hospital, Ludhiana
  - Department of Medical Oncology, Jaslok Hospital and Research Centre, Mumbai
- Poland (6):
  - Colorectal Cancer Clinic, Centrum Cancer Clinic Onkologii-Instytut im M. Skladowskiej-Curie, Roentgena, Warszawa
  - Department and Clinic for Oncology and Radiotherapy, Gdansk
  - Department for Oncology and Radiotherapy, Szpital Morski im. PCK, Gdynia Redlowo
  - Oncological Chemotherapy Clinic, Regionalny Osrodek Onkologiczny, Lodz
  - Oncological Chemotherapy Department Centrum Onkologii Ziemi, Lublin
  - Clinical Oncology Department, Wojewodski Szpital Zespolony, Torun
- Romania (4):
  - Gastroenterology and Hepatology Department, Fundeni Clinical Institute, Bucharest
  - Professor of Dr. Alexandru Trestioreanu, Institute of Oncology II, Bucharest
  - Department of Medical Oncology and Radiotherapy II, Cluj-Napoca
  - Medical Oncology Department, County Hospital Sibiu, Sibiu
- Serbia (7):
  - Clinical Center of Serbia, Belgrade
  - Institute of Oncology and Radiology Serbia, Belgrade
  - CHC Bezanijska, Belgrade
  - Clinic for Internal Medicine, Institute for Oncology Sremska, Kamenitz
  - CHC Kragujevac, Kragujevac
  - Clinic Centre Nis, Niš
  - General Hospital Djordje Joanovic, Zrenjanin
- United Kingdom (3):
  - Haematology/Lung/GI Cancer Services, Harlow, Essex
  - Oncology Research, North Middlesex University Hospital, Middlesex, London
  - Beatson Oncology Centre, Glasgow